CLINICAL TRIAL: NCT01413815
Title: Effect of Oral Supplementation With the Amino Acid L-arginine on Peri- Operative Cardio-vascular Risk in Non-selected Patients - Role of Pre-operative Determination of Plasma ADMA Levels for Therapeutic Stratification.
Brief Title: Effect of the Amino Acid L-arginine on Perioperative Cardio-vascular Risk in Non-selected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UKE-KP 2009/001
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Cardiovascular Complication
Keywords: peri-operative; cardiovascular risk; oral supplementation; amino acid L-arginine
MeSH Terms: interventions — Arginine; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-arginine (Active Comparator): L-Arginine
  Interventions: Dietary Supplement: L-arginine
- corn starch (Placebo Comparator): Placebo: Corn Starch
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: L-arginine — 3.3 g of L-arginine capsules, oral,b.i.d for a period of three days (a variability ±2 days is accepted to enable scheduling of surgery according to requirements of clinical routine).
  Arms: L-arginine
Other: Placebo — 3.3 g of placebo capsules/ b.i.d.; for a period of three days (a variability ±2 days is accepted to enable scheduling of surgery according to requirements of clinical routine)
  Other Names: corn starch
  Arms: corn starch

SUMMARY:
The aim of the study is to test whether pre-operative oral supplementation with L-arginine results in a significant reduction of peri-operative cardiovascular complication rate in unselected patients undergoing major abdominal or thoracic (non-cardiac) surgery. The second aim of the study is to assess whether pre-operative determination of plasma ADMA levels allows to identify patients who are at high risk of experiencing a peri-operative complication, and whether this subgroup of patients profits specifically from pre-operative L-arginine supplementation.

DETAILED DESCRIPTION:
Patients will be recruited for this study from the participating Departments. In a previous study (protocol no. UKE-KP 2002/006) we investigated the predictive role of ADMA (asymmetric dimethylarginine) for peri-operative complications in unselected patients undergoing major surgery. The major result of that study was that patients with pre-operative ADMA plasma level within the highest quartile of the distribution had a significantly elevated risk of experiencing a serious peri-operative complication within a period of 30 days after the surgical intervention. These data have been published [Maas et al. 2007]. As ADMA competitively displaces L-arginine from the enzyme, NO synthase, it is expected that the adverse cardiovascular effects of high ADMA levels can be antagonized by supplemental L-arginine. Therefore, the present study was designed to specifically address the question whether dietary supplementation with L-arginine before the surgery, aiming at replenishing the body's L-arginine stores, may help to reduce the peri- operative complication rate. Another aim is to assess whether this occurs in all patients or specifically in the subgroup with elevated baseline ADMA levels.

Study participants will be recruited from patients who routinely visit the outpatient clinic at the participating Departments of Anesthesiology and Intensive Care in advance of their planned surgical intervention. Patients usually visit the clinic between five working days in advance of the scheduled time of surgery, or they are admitted to in-patient treatment one or two days before the surgery. They will be informed about the scope and aim of the study, and after having given their informed consent, patients will receive L-arginine dietary supplements or corresponding placebo according to randomisation plan for the time until surgery. The last dosage of the L-arginine supplements will be taken in the morning of the surgery, dissolved in a glass of tap water that patients ware required to drink with premedication for anesthesia. Blood samples to measure plasma L-arginine and ADMA levels will be taken at the time of inclusion, in the morning before scheduled surgery, and on days 1 and 3 after the surgery and will together with additional safety parameter not exceed 80ml. No administration of study product will occur after surgery.

After surgery having taken place, patients will be monitored daily for as long as they remain being treated as in-patients, and all clinical events, changes in laboratory parameters, and apparatively performed clinical tests as scheduled according to clinical routine will be documented. No additional clinical treating will be performed on study participants, except the blood samples that will be taken as described above. After discharge, patients will be followed-up telephonically, for the last time at 30 days after the date of surgery. All clinical events occurring in this period will be recorded. In addition, changes in laboratory values, ECG recordings, and other apparative diagnostic measures will be checked for possible complications, and also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects aged between 30 and 75 years;
* scheduled major thoracic (non-cardiac), abdominal, or two cavity surgery;
* ASA risk class II- IV;
* efficient birth control for women in child-bearing age;
* signed written informed consent form.

Exclusion Criteria:

* participation in a clinical study within the last 3 months before inclusion into the present study;
* high allergic tendency in the medical history at the investigators discretion;
* patients with known diabetic retinopathy;
* previous abuse of drugs or alcohol;
* pregnancy or nursing;
* any severe consuming disease (malignant or non-malignant) that reduces the patient's life expectancy to a level which makes it uncertain that the patient would survive the 30 day period even without surgery;
* any somatic or psychic disease that may hamper participation in the study or compliance;
* active liver disease or hepatic failure (serum AST or ALT >1.5-fold above the upper limit of the normal range);
* severe renal failure (calculated creatinine clearance < 30 ml/min [Cockcroft-Gault formula]), nephrotic syndrome or dysproteinemia;
* previous intolerance of L-arginine or L-citrulline.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2010-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
difference in incidence of the combined end-point of death of any cause | period of 30 days after surgery
  the difference in incidence of the combined end-point of death of any cause, acute myocardial infarction or acute coronary syndrome, decompensated heart failure, cardiac arrest or resuscitation, and cerebral or pulmonary embolism between L-arginine and placebo.

SECONDARY OUTCOMES:
difference in incidence between L-arginine and placebo (subgroup with ADMA) | period of 30 days after surgery
  difference in incidence between L-arginine and placebo for the subgroups with ADMA below and above the median concentration
difference in incidence between beta-blocker or no beta-blocker treatment | period of 30 days after surgery
  the difference in incidence of the combined primary end-point between patients on beta-blocker treatment or not on beta-blocker treatment
difference in incidence between statin treatment or no statine treatment | period of 30 days after surgery
  the difference in incidence of the combined primary end-point between patients on statin treatment or not on statin treatment
difference in incidence between L-arginine and placebo (ASA class) | period of 30 days after surgery
  -the difference in incidence of the combined primary end-point between L-arginine and placebo for each of the ASA classes II to IV

CONTACTS AND LOCATIONS:
Overall Officials: Rainer H. Böger, Professor, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (5):
- Germany (5):
  - Klinik für Anästhesiologie,Städtisches Klinikum Lüneburg, Lüneburg, Lower Saxony
  - Institut für Experimentelle und Klinische Pharmakologie,Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Klinik für Anästhesiologie, Intensivmedizin und Schmerztherapie,Kath. Marienkrankenhaus gGmbH, Hamburg
  - Klinik und Poliklinik für Anästhesiologie, Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Klinik für Anästhesie und operative Intensivmedizin,Asklepios Klinik Nord, Standort Heidberg, Hamburg

REFERENCES:
- [Background] Maas R, Dentz L, Schwedhelm E, Thoms W, Kuss O, Hiltmeyer N, Haddad M, Kloss T, Standl T, Boger RH. Elevated plasma concentrations of the endogenous nitric oxide synthase inhibitor asymmetric dimethylarginine predict adverse events in patients undergoing noncardiac surgery. Crit Care Med. 2007 Aug;35(8):1876-81. doi: 10.1097/01.CCM.0000277038.11630.71. PMID 17581491
- [Result] Appel D, Boger R, Windolph J, Heinze G, Goetz AE, Hannemann J. Asymmetric dimethylarginine predicts perioperative cardiovascular complications in patients undergoing medium-to-high risk non-cardiac surgery. J Int Med Res. 2020 Aug;48(8):300060520940450. doi: 10.1177/0300060520940450. PMID 32842812